CLINICAL TRIAL: NCT00472901
Title: A Phase III, Randomised, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of Subcutaneous Implants of CUV1647 in Patients Suffering From Polymorphic Light Eruption (PLE).
Brief Title: Phase III Trial of CUV1647 in Polymorphic Light Eruption (PLE)
Status: Completed | Type: Observational
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CUV015
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Polymorphic Light Eruption (PLE)
Keywords: Polymorphic Light Eruption (PLE); Afamelanotide; CUV1647; photoprotection; sun poisoning
MeSH Terms: interventions — afamelanotide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Afamelanotide (CUV1647) — 16mg implant

SUMMARY:
The purpose of this study is to determine whether the afamelanotide (CUV1647) formulation is effective in preventing PLE episodes or reducing the severity of PLE symptoms in patients with a well documented history of the disease. The study also aims to determine whether treatment with afamelanotide (CUV1647) can reduce the use of rescue medication in this group.

DETAILED DESCRIPTION:
Polymorphic Light Eruption (PLE) is a prevalent photosensitivity disorder, occurring in up to 20% of the European and US populations and up to 5% of the Australian population. The disease is characterised by a rash that is intensely itchy with blisters, bumps and patches presenting on areas of the skin that have been exposed to the sun. There is a lack of effective treatment available for the condition but the most common available forms of therapy include sun avoidance and the use of the use of steroids and/or phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 70 years at inclusion.
* Well documented history of moderate/severe PLE as diagnosed/confirmed by a photodermatologist or photobiologist. Newly diagnosed patients with moderate/severe PLE can be included if numbers of established patients are limited provided their diagnosis is confirmed by a photodermatologist or photobiologist.
* Recurrent episodes that occur at least once a year, developing in own country (to exclude patients affected only when traveling to sunnier climates).
* Have given written informed consent to participate in the study.

Exclusion Criteria:

* Personal history of melanoma, lentigo maligna or multiple (3 or more) dysplastic nevi.
* Current Bowen's Disease, basal cell carcinoma, squamous cell carcinoma or other malignant skin lesions.
* Documented history of other photosensitive conditions.
* Female who is pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating.
* Females of child-bearing potential that are not using adequate contraceptive measures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate/severe polymorphic light eruption (PLE)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate whether afamelanotide (CUV1647) prevents episodes or reduces the severity of PLE symptoms in patients with a well documented history of PLE | 18 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of afamelanotide (CUV1647) in this specific clinical setting | 18 months
To evaluate the effect of afamelanotide (CUV1647) on melanin density levels as measured by skin reflectance | 18 months
To evaluate whether afamelanotide (CUV1647) has a beneficial effect on the quality of life of patients with a documented history of PLE | 18 months
To determine if there are other factors that may influence the severity of PLE symptoms eg. sun exposure and use of sun protection methods | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Rhodes, MD, Principal Investigator — Hope Hospital, Manchester, United Kingdom; Herbert Hoenigsmann, MD, Principal Investigator — Medical University of Vienna; Chris Baker, MD, Principal Investigator — St. Vincent's Hospital, Melbourne, AUSTRALIA
Locations (3):
- St Vincents Hospital, Melbourne, Australia
- Medical University of Vienna, Vienna, Austria
- Hope Hospital, Manchester, United Kingdom